CLINICAL TRIAL: NCT00517777
Title: Effects of the Continuous Positive Airway Pressure Ventilation on the Prevalence of the Metabolic Syndrome and Cardiac Morpho-Functional Characteristics in Sleep Apnea Syndrome
Brief Title: Continuous Positive Airway Pressure in Sleep Apnea Syndrome: Effects on Metabolic Syndrome and Cardiac Damage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1113
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Sleep Apnea Syndrome; Metabolic Syndrome; Cardiac Remodelling; Continuous Positive Airway Pressure Ventilation
Keywords: sleep apnea syndrome; metabolic syndrome; cardiac remodelling; continuous positive airway pressure ventilation
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Syndrome | interventions — Continuous Positive Airway Pressure; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): continuous positive airway pressure ventilation + dietary and life style recommendations
  Interventions: Device: continuous positive airway pressure ventilation; Behavioral: dietary and life style recommendations
- 2 (Active Comparator): dietary and life style recommendations
  Interventions: Behavioral: dietary and life style recommendations

INTERVENTIONS:
Device: continuous positive airway pressure ventilation — nighttime
  Arms: 1
Behavioral: dietary and life style recommendations
  Arms: 2
Behavioral: dietary and life style recommendations
  Arms: 1

SUMMARY:
To assess in moderate to severe Obstructive Sleep Apnea the effects of one year therapy with nighttime continuous positive airway pressure ventilation on the prevalence of metabolic syndrome and cardiovascular damage.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe sleep apnea syndrome

Exclusion Criteria:

* cardiovascular diseases (coronary artery disease, stroke, peripheral artery disease)
* thyroid diseases
* diabetes

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
metabolic syndrome | one year
left ventricular mass | one year
diastolic function | one year

CONTACTS AND LOCATIONS:
Overall Officials: anna maria grandi, MD, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- University of Insubria-Department of Clinical Medicine, Varese, Italy

REFERENCES:
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; American Heart Association; National Heart, Lung, and Blood Institute. Definition of metabolic syndrome: Report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Circulation. 2004 Jan 27;109(3):433-8. doi: 10.1161/01.CIR.0000111245.75752.C6. No abstract available. PMID 14744958
- [Background] Cloward TV, Walker JM, Farney RJ, Anderson JL. Left ventricular hypertrophy is a common echocardiographic abnormality in severe obstructive sleep apnea and reverses with nasal continuous positive airway pressure. Chest. 2003 Aug;124(2):594-601. doi: 10.1378/chest.124.2.594. PMID 12907548
- [Background] Norman D, Loredo JS, Nelesen RA, Ancoli-Israel S, Mills PJ, Ziegler MG, Dimsdale JE. Effects of continuous positive airway pressure versus supplemental oxygen on 24-hour ambulatory blood pressure. Hypertension. 2006 May;47(5):840-5. doi: 10.1161/01.HYP.0000217128.41284.78. Epub 2006 Apr 3. PMID 16585412
- [Background] Shivalkar B, Van de Heyning C, Kerremans M, Rinkevich D, Verbraecken J, De Backer W, Vrints C. Obstructive sleep apnea syndrome: more insights on structural and functional cardiac alterations, and the effects of treatment with continuous positive airway pressure. J Am Coll Cardiol. 2006 Apr 4;47(7):1433-9. doi: 10.1016/j.jacc.2005.11.054. Epub 2006 Mar 15. PMID 16580533